CLINICAL TRIAL: NCT05671146
Title: An Evaluation of the Graded Weight-bearing Exercise on Pain, Function, Proprioception, and Muscle Strengths in Patients With Knee Osteoarthritis.
Brief Title: An Evaluation of the Graded Weight-bearing Exercise in Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ammar Fadil, Principle Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-PGS-2022-03-447
Record Dates: First submitted 2022-12-07; First posted 2023-01-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
Keywords: Graded weight-bearing exercise; Anti-gravity treadmill
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: knee osteoarthritis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Graded weight-bearing exercise (Experimental): participants will perform exercises using an anti-gravity treadmill
  Interventions: Device: anti-gravity treadmill
- Closed kinetic chain exercise (Active Comparator): Exercises will be achieved in a weight-bearing position, with or without support, besides other exercises to improve knee flexors and extensors strength.
  Interventions: Other: Weight-bearing exercises for knee flexors and extensors
- open kinetic chain exercise (Sham Comparator): Exercises including stretching and strengthening exercises for knee flexors and extensors
  Interventions: Other: Non weight-bearing exercises for knee flexors and extensors

INTERVENTIONS:
Device: anti-gravity treadmill — participants will perform exercises with partial weight-bearing by using an anti-gravity treadmill
  Arms: Graded weight-bearing exercise
Other: Weight-bearing exercises for knee flexors and extensors — Stretching and strengthening exercises will be performed in a weight-bearing position
  Arms: Closed kinetic chain exercise
Other: Non weight-bearing exercises for knee flexors and extensors — Stretching and strengthening exercises will be performed in a non-weight-bearing position
  Arms: open kinetic chain exercise

SUMMARY:
Background: Knee osteoarthritis is the most common disorder impacting the synovial joint. The prevalence of osteoarthritis rises with age, and its consequences on health and socioeconomic are significant, which emphasize the need for clinical and cost-effective treatments for patients with knee OA. Knee OA is a widespread joint arthritis disease combined with many clinical features such as pain, decreased joint proprioception and might lead to loss of function and disability.

Aim: To evaluate the effect of a 6-weeks supervised graded weight-bearing exercise program on pain, function, proprioception, muscle strength in patients with knee osteoarthritis.

Material and Method: Thirty-six patients with chronic knee osteoarthritis with age ranging 40-60 years will be recruited from the physical therapy department and randomized into three groups. Group I: will receive graded weight-bearing exercise using the anti-gravity treadmill combined with open kinetic chain exercises. Group II will receive closed kinetic chain exercises with open kinetic chain exercises while group III will receive open kinetic chain exercises only i.e: stretching and strengthening exercises. The outcome measures will be pain, function, proprioception, and muscle strength.

Statistical analysis: To detect changes in the dependent variables within and between groups, one-way repeated measures Multivariate analysis will be applied. If there is a significant change within groups or between tests, the post hoc Bonferroni test will be used to detect the significance between each group and/or each level of measurement. The level of significance is p<0.05 and confidence interval CI 95%.

Study Design: Single-blinded, randomised control trial.

DETAILED DESCRIPTION:
Study design: This study is a single-blinded randomized controlled trial. after baseline assessment, the participants will be assigned randomly into three groups, the graded weight-bearing exercise group, the closed kinetic chain exercise group, and the control group. First, randomization will be performed by allocating a specific number for each participant. Then, Online GraphPad will be applied to randomize these numbers into three groups. The participants' allocation will be conducted by a person who is not in contact with the participants or involved in any testing. The allocation sequence will be saved on that person's computer. Following randomization, the participant will be notified by phone about which group they will be assigned to.

Study setting: The current study will be held at the laboratory at Umm Al-Qura University, Faculty of Applied Medical Sciences, Makkah, Saudi Arabia Recruitment and study population Patients will be recruited from the physical therapy outpatient clinic, Umm Al-Qura university medical centre, and other physical therapy outpatient clinic in Makkah.

Intervention group:

The intervention will be constructed based on recent clinical exercise guidelines for people with knee osteoarthritis. These guidelines mainly recommend weight-bearing exercises, progressive resistance training for lower limb major muscle groups, and aerobic exercise. The exercise regimen will be applied at two sessions per week for six weeks. The intervention is designed as the group I will perform progressive weight-bearing using an anti-gravity treadmill, the loading starts with patient tolerance - pain-free range and increases gradually, combined with open kinetic chain exercises. Group II will perform closed kinetic chain exercises with open kinetic chain exercises. Most of the exercises in these groups will be achieved in a weight-bearing position, with or without support, besides other exercises to improve knee flexors and extensors strength. An experienced physiotherapist will observe the intervention. Participants who have a higher risk of falling, restricted weight-bearing activities, or movement during training and activities will be given extra attention to avoid injuries. The physiotherapists will be trained to deliver the weight-bearing exercise program and ensure that participants have access to support devices. The session will last one hour and be repeated twice a week for six weeks. Participants' customizing, appropriate dosage, and progression of the exercises will be the responsibility of the physiotherapist supervising the exercise session. The exercise regimen will begin with a 10-minute warm-up that includes stretching, flexibility, and dynamic balance exercises. The warm-up will be followed by a graded weight-bearing exercise for group I and a closed kinetic chain exercise for group II with a short break for 30 seconds. Each session will end with 10 min cooling down and stretching. Participants are encouraged to report any significant side effects from the exercise, such as muscular soreness, joint tenderness, or increased pain level.

Control group:

Participants assigned to the control group will receive open kinetic chain exercises only, including stretching and strengthening exercises for knee flexors and extensors. They will be expected to maintain their current level of physical activity and go about their daily lives as usual.

Adherence:

The percentage of total intervention days completed will be used to determine adherence. 12 sessions = 100%.

Sample size estimation: A G-power grogram for windows is used to calculate the estimated sample size with an effect size of 0.25 and an alpha error probability of 0.90 to detect the changes in three groups receiving three independent interventions for four dependent variables. The measurement will be repeated twice across the study period. The statistical test used is the Multivariate Analysis of variance (MANOVA), and the total sample size will be 36. The number will be increased for possible dropout to 45 patients with 15 patients in each group. Statistical Analysis The study's findings will be presented in accordance with CONSORT.

Statistical analysis: will be carried out with the help of statistical software such as SPSS. Patients' demographic data will be presented as mean and standard deviation. Analysis of the patients' age (years), weight (Kg), height (cm), and body mass index (BMI) kg/m2 will be performed by one-way analysis of variance (ANOVA) to detect the similarity in subjects between the treatment groups. Three treatment groups that received three different interventions will be measured twice at pre-treatment and post-treatment. To detect changes in the dependent variables within and between groups, one-way repeated measures Multivariate analysis (MANOVA) will be applied. If there is a significant change within groups or between tests, the post hoc Bonferroni test will be used to detect the significance between each group and/or each level of measurement. The level of significance is p<0.05. The data will be analyzed with the intention to treat principles. Each paper from the project will be subjected to a statistical analysis publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients had chronic pain in either unilateral or bilateral knees ≥ 6 months.
* The x-ray showed grades II and III according to on Kallgren and Lawrence (K/L) grading system.
* Patients are willing to stop medications.
* Patients accepted to assign informed consent to participate in the current study and will attend the lab twice a week for six successive weeks.

Exclusion Criteria:

* They have any known significant medical conditions such as hypertension, asthma, cardiac disease, or systemic disease that adversely affect them during testing.
* Previous knee surgery/injection for the last six months.
* Previous knee fracture or malignancy.
* Unable to walk unaided.
* Unable to commit study requirements.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Measurment of pain intensity | Change from Baseline Pain Intensity at 6 weeks post-intervention
  The pain will be measured using a visual analogue scale (VAS). This scale is a 10-centimeter drawn line. Zero indicates no pain or discomfort, and 10 indicates the most severe pain. The patient will be asked to mark on the line corresponding to their pain level. For patients with chronic musculoskeletal pain, the VAS is a valid and reliable measure.
Function | Change from Baseline Functional level at 6 weeks post-intervention
  The function will be measured by WOMAC. The WOMAC index is a sensitive, validated, and reliable measure of knee osteoarthritis impacts such as functional conditions. The WOMAC scale has 17 items used to assess patients with osteoarthritis physical function. The patient's response runs from 1 to 5, with 1 indicating no response and 5 indicating a strong response. The total score will be calculated by adding the scores for each item.

SECONDARY OUTCOMES:
Proprioception | Change from Baseline Knee Joint Proprioception at 6 weeks post-intervention
  The proprioception will be measured using the joint position sense method. The Biodex System isokinetic dynamometer is a reliable apparatus for measuring angular joint position.
Muscle strength | Change from Baseline Quadriceps Muscles strength at 6 weeks post-intervention
  The dynamometer is a proven and accurate way to assess quadriceps muscle strength. To control the effects of fatigue, the strength testing was done in the order of 120°/s, 180°/s, and finally 60°/s. On the testing side, participants are set leaning against a backrest tilted 15 degrees backward from vertical and will be strapped to the machine at the upper chest, pelvis, and distal femur. The participants will be instructed to extend their knee as far as possible, with the highest values from the three trials recorded as peak torque at each speed. The gravity of all data will be rectified.

CONTACTS AND LOCATIONS:
Overall Officials: Ammar S Fadil, Ph.D, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- Umm Al-Qura University, Mecca, Western Chapter, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No